CLINICAL TRIAL: NCT04059679
Title: Synergistic Influence of Rivaroxaban on Inflammation and Coagulation Biomarkers in Patients With CAD and PAD on Aspirin Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LifeBridge Health (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1436289
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Coronary Artery Disease; Peripheral Artery Disease
MeSH Terms: conditions — Coronary Artery Disease; Peripheral Arterial Disease | interventions — Rivaroxaban; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EC aspirin (81mg qd) (Active Comparator)
  Interventions: Drug: Aspirin 81 mg
- EC aspirin (81mg qd) plus rivaroxaban (2.5 mg bid) (Experimental)
  Interventions: Drug: Rivaroxaban 2.5 Mg Oral Tablet; Drug: Aspirin 81 mg

INTERVENTIONS:
Drug: Rivaroxaban 2.5 Mg Oral Tablet — EC aspirin (81mg qd) plus rivaroxaban (2.5 mg bid)
  Arms: EC aspirin (81mg qd) plus rivaroxaban (2.5 mg bid)
Drug: Aspirin 81 mg — EC aspirin 81 mg qd

SUMMARY:
This is a phase IV, prospective biomarker study that will be conducted at Sinai Hospital of Baltimore. After screening for patients who were treated with aspirin, thirty patients will be treated with 81 mg enteric coated (EC) aspirin for 7 days in the "lead-in" period and then will be randomly treated with EC aspirin (81mg qd) or EC aspirin (81mg qd) plus rivaroxaban (2.5 mg bid) for 12 weeks. Platelet aggregation, soluble markers of platelet activation and inflammation, thrombin generation kinetics and tissue factor (TF)-induced platelet-fibrin clot strength will be assessed at baseline (after 7 days of treatment with 81 mg EC aspirin), and 4 and 12 weeks after randomization of the study drug administration.

ELIGIBILITY:
Inclusion Criteria: to qualify, all subjects must meet have CAD and PAD as according to criteria specified below:

* Subjects meeting criteria for CAD$ must have one or more of the following:
* Myocardial infarction within the past 20 years, or
* Multivessel coronary disease* with symptoms or with history of stable or unstable angina, or
* Multivessel percutaneous coronary intervention, or
* Multivessel CABG surgery (* Refers to stenosis of ≥ 50% in 2 or more coronary arteries, confirmed using invasive coronary angiography, or noninvasive imaging or stress studies (eg, exercise or pharmacologic) suggestive of significant ischemia in 2 ≥ coronary territories; or in 1 coronary territory if at least 1 other territory has been revascularized.)

$Subjects with the qualifying criteria of CAD must also met at least one of the following criteria:

* Age > 65 years, or
* Age <65 years and documented atherosclerosis or revascularization involving at least 2 vascular beds+, or at least 2 additional cardiovascular risk factors:

  1. Current smoker (within 1 year of randomization)
  2. Diabetes mellitus
  3. Renal dysfunction with estimated glomerular filtration rate of <60 ml/min
  4. Heart failure
  5. Non-lacunar ischemic stroke > 1 month ago

     * Because CAD involves disease in the coronary vasculature, only one additional vascular bed is required: e.g. the aorta and arterial supply to the brain, gastro-intestinal tract, lower limbs, upper limbs, or kidneys.

       * Subjects meeting criteria for PAD must have one or more of the following
* Previous aorto-femoral bypass surgery, limb bypass surgery, or percutaneous transluminal angioplasty revascularization of the iliac, or infrainguinal arteries, or
* Previous limb or foot amputation for arterial vascular disease (i.e., excludes trauma), or
* History of intermittent claudication and one of the following

  * An ankle/arm blood pressure (BP) ratio < 0.90,
  * Significant peripheral artery or venous stenosis of ≥50% documented by angiography or by duplex ultrasound
  * Previous carotid revascularization or asymptomatic carotid artery stenosis ≥ 50% as diagnosed using duplex ultrasound or angiography.

    * Subject may be of either sex and of any race, and must be >18 years of age.
    * Subject agrees to not participate in any other investigational or invasive clinical study for a period of 4 months during the study period
    * The subject is able to read and has signed and dated the informed consent document including authorization permitting release of personal health information approved by the investigator's Institutional Review Board (IRB).

Exclusion Criteria: Subjects will be excluded from entry if ANY of the criteria listed below are met:

* High risk of bleeding
* Stroke within 1 month or any history of hemorrhagic or lacunar stroke
* Severe heart failure with known ejection fraction <30% or New York Heart Association (NYHA) class III or IV symptoms
* Estimated glomerular filtration rate (eGFR)<15 mL/min
* Need for dual antiplatelet therapy, other non-aspirin antiplatelet therapy, or oral anticoagulant therapy
* Known non-cardiovascular disease that is associated with poor prognosis (e.g., metastatic cancer) or that increases the risk of an adverse reaction to study interventions.
* History of hypersensitivity or known contraindication for rivaroxaban, aspirin, or its excipients. Systemic treatment with strong inhibitors of both CYP 3A4 and p-glycoprotein (P-gp) (e.g., systemic azole antimycotics, such as ketoconazole, and human immunodeficiency virus [HIV]-protease inhibitors, such as ritonavir), or strong inducers of CYP 3A4, i.e. rifampicin, rifabutin, phenobarbital, phenytoin, and carbamazepine.
* Participation in any investigational study within the last 60 days.
* Active liver disease or hepatic dysfunction, defined as AST or ALT >3 x ULN as determined by laboratory test results drawn at or available during screening.
* Recipient of any major organ transplant (e.g., lung, liver, heart, bone marrow, renal).
* Subjects with prosthetic heart valves.
* Known major active infection or major hematologic, renal, metabolic, gastrointestinal, or endocrine dysfunction in the judgment of the investigator.
* Malignancy (except non-melanoma skin cancers, cervical in situ carcinoma, breast ductal carcinoma in situ, or stage 1 prostate carcinoma) within the last 5 years.
* Subject is pregnant or breast feeding, or planning to become pregnant or to breastfeed during receipt of investigational products and within 15 weeks after the end of study treatment.
* Female subject who is unwilling to use at least 2 effective birth control methods for at least 1 month before screening and 15 weeks after the end of treatment with investigational products, unless the subject is sterilized or postmenopausal.
* Subject likely to not be available to complete all protocol-required study visits or procedures, to the best of the subject's and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition, or disease other than those outlined above that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Relative Difference in maximal ADP-induced Platelet Aggregation | 12 weeks
  Relative difference in maximal ADP-induced platelet aggregation between 81mg qd EC aspirin or 81mg qd EC aspirin plus 2.5 mg bid rivaroxaban therapy for 12 weeks.

SECONDARY OUTCOMES:
Relative differences in TF-thrombin-induced platelet aggregation | 12 weeks
  Relative differences in TF-thrombin-induced platelet aggregation between 81mg qd EC aspirin or 81mg qd EC aspirin plus 2.5 mg bid rivaroxaban therapy for 12 weeks.
Relative differences in alpha- thrombin-induced platelet aggregation | 12 weeks
  Relative differences in alpha- thrombin-induced platelet aggregation between 81mg qd EC aspirin or 81mg qd EC aspirin plus 2.5 mg bid rivaroxaban therapy for 12 weeks.
Relative differences in inflammation biomarkers | 12 weeks
  Relative differences in IL-6, hsCRP, platelet bound p-selectin, VCAM, fibrinogen, oxLDL, oxLDL/atherox, TAT complexes, prothrombin F1+2, D-dimer and FpA (soluble markers) between 81mg qd EC aspirin or 81mg qd EC aspirin plus 2.5 mg bid rivaroxaban therapy for 12 weeks
Relative differences in platelet-fibrin clot characteristics | 12 weeks
  Relative differences in platelet-fibrin clot characteristics between 81mg qd EC aspirin or 81mg qd EC aspirin plus 2.5 mg bid rivaroxaban therapy for 12 weeks
Relative differences in shear-induced platelet aggregation | 12 weeks
  Relative differences in shear-induced platelet aggregation between 81mg qd EC aspirin or 81mg qd EC aspirin plus 2.5 mg bid rivaroxaban therapy for 12 weeks
Relative differences in lag time | 12 weeks
  Relative differences in lag time between 81mg qd EC aspirin or 81mg qd EC aspirin plus 2.5 mg bid rivaroxaban therapy for 12 weeks
Relative differences in peak thrombin production | 12 weeks
  Relative differences in peak thrombin production between 81mg qd EC aspirin or 81mg qd EC aspirin plus 2.5 mg bid rivaroxaban therapy for 12 weeks
Relative differences in mean velocity rate index | 12 weeks
  Relative differences in mean velocity rate index between 81mg qd EC aspirin or 81mg qd EC aspirin plus 2.5 mg bid rivaroxaban therapy for 12 weeks
Relative differences in endogenous thrombin potential | 12 weeks
  Relative differences in endogenous thrombin potential between 81mg qd EC aspirin or 81mg qd EC aspirin plus 2.5 mg bid rivaroxaban therapy for 12 weeks

OTHER OUTCOMES:
First occurrence of modified ISTH major bleeding | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sinai Hospital of Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tantry U, Cummings C, Mackrell P, Gonze M, Ulloa K, Bafford R, Rout A, Sukhi A, Gurbel P. Synergistic influence of rivaroxaban on inflammation and coagulation biomarkers in patients with coronary artery disease and peripheral artery disease on aspirin therapy. Future Cardiol. 2020 Mar;16(2):69-75. doi: 10.2217/fca-2019-0091. Epub 2020 Mar 4. PMID 32129681